CLINICAL TRIAL: NCT02903238
Title: Brain Morphometric Study in Knee Osteoarthritis Patients Treated With Duloxetine
Brief Title: Brain Morphometry in OA Patients Treated With Duloxetine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Apkar Apkarian, Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: STU00039556A
Record Dates: First submitted 2016-08-26; First posted 2016-09-16 (Estimated); Results first posted 2017-03-07 (Actual); Last update posted 2017-03-07 (Actual); Status verified 2017-01

CONDITIONS: Pain; Osteoarthritis
Keywords: placebo; pain; osteoarthritis
MeSH Terms: conditions — Pain; Osteoarthritis | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Placebo (Experimental): placebo capsule
  Interventions: Drug: Duloxetine; Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Duloxetine — Duloxetine Delayed-Release Capsules: 30mg/day for 1 week ; 60mg/day for the remaining time
  Other Names: Cymbalta
Drug: Placebo Oral Tablet — Lactose capsule
  Other Names: Placebo

SUMMARY:
This is a two week,single-blind study evaluating pain response and changes in brain imaging upon treatment with placebo in people with knee OA.

DETAILED DESCRIPTION:
In this study, all the participants will be receiving placebo. However this study will be single blinded in that participants will be told that they will be given a pill that may or may not help with their pain. The researcher, however, will know that all participants are receiving placebo

At the initial visit, participants will undergo screening to determine that they meet all inclusion and exclusion criteria. They will sign consent and then complete pain assessment instruments as well as one high resolution anatomical scan (T1) and one functional scan (a resting scar) in a 3 Tesla magnet. A single scanning session comprised of a 10 minute functional scan (a resting scan) will be done two weeks from the first scan and pain assessment instruments will be completed at this visit as well. After finishing this second scan (done two weeks after the initial scan), the participants will have completed the study.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40-85 years
* ACR criteria for OA including Kellgren-Lawrence radiographic OA grades II-IV
* VAS pain score >5/10 within 48 hrs of the phone screen and visit 1 (Screening)
* Knee OA for a minimum of 12 months
* Need for daily pain medication to manage symptoms of OA

Exclusion Criteria:

* Currently taking MAO inhibitors or any centrally acting drug for analgesia
* Narrow angle glaucoma
* Uncontrolled hypertension
* Co-existing inflammatory arthritis, fibromyalgia or other chronic pain state
* If a female, pregnant, trying to become pregnant, or lactating
* Major depressive disorder
* Substantial alcohol use or history of significant liver disease
* Diabetes, type 1 or type 2
* Condition in which the Investigator believes would interfere with the subject's ability to comply with study instructions, or might confound the interpretation of the study results or put the subject at undue risk
* Standard MRI safety exclusions

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-07; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Apkar V Apkarian, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
The data will be available at http://OpenfMRI.org

REFERENCES:
- [Derived] Tetreault P, Mansour A, Vachon-Presseau E, Schnitzer TJ, Apkarian AV, Baliki MN. Brain Connectivity Predicts Placebo Response across Chronic Pain Clinical Trials. PLoS Biol. 2016 Oct 27;14(10):e1002570. doi: 10.1371/journal.pbio.1002570. eCollection 2016 Oct. PMID 27788130

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: placebo capsule
  placebo: lactose containing capsule
Period: Overall Study
Arm/Group | Placebo
Started | 21
Completed | 17
Not Completed | 4
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | Placebo
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.88 (5.68)
Gender [Count of Participants; unit: Participants]
  Female | 9
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 17
Pain (Visual Analogue Score, VAS) [Mean (Standard Deviation); unit: units on a scale] — 0 to 10 (0=no pain, 10=worst pain)
  units on a scale | 7.03 (1.08)

OUTCOME MEASURES:

1. Primary Outcome: Brain Regional Gray Matter Density
Description: Gray matter density (GMD) of the prefrontal cortex region identified as placebo biomarker. Placebo responders/non-responders were identified based on the VAS score. A minimum of 20% decrease in VAS score was needed to be qualified as responders.
  GMD is a value between 0 and 1 representing the intensity of every brain voxels. The GMD of the prefrontal cortex region represent the average GMD of every voxels in this region.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: Gray Matter Density: 0 to 1
Groups:
- Placebo Responders; Placebo Non-responders: placebo capsule
  placebo: lactose containing capsule
Arm/Group | Placebo Responders | Placebo Non-responders
Number analyzed (Participants) | 8 | 9
Gray Matter Density: 0 to 1 | 0.420 (0.083) | 0.425 (0.060)

2. Secondary Outcome: WOMAC Pain Index
Description: Osteoarthritis (OA) specific pain and quality of life index (the Western Ontario and McMaster Universities Osteoarthritis Index WOMAC). The WOMAC score is from 0 to 96 where 0 represent no pain and quality of life impairment due to OA and 96 represent the worst pain and quality of life impairment due to OA. The outcome is reported as the percent change from baseline to end of treatment (2 weeks).
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: Percent Change in WOMAC score
Arm/Group | Placebo Responders | Placebo Non-responders
Number analyzed (Participants) | 8 | 9
Percent Change in WOMAC score | 38.6 (24.6) | 4.6 (21.3)

3. Secondary Outcome: Overall Brain Neocortical Gray Matter Volume
Time Frame: 2 weeks
Population: Data were not collected and the Outcome will never be analyzed
Arm/Group | Placebo Responders | Placebo Non-responders
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Placebo
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No